CLINICAL TRIAL: NCT03806491
Title: The Impact of CBT for Insomnia on Alcohol Treatment Outcomes Among Veterans
Brief Title: CBT-I on Alcohol Treatment Outcomes Among Veterans
Acronym: Project SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Harry S. Truman Memorial Veterans' Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary E Miller, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012262
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Insomnia; Alcohol Use Disorder
Keywords: veteran; alcohol; insomnia; sleep; drinking
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcoholism | interventions — Cognitive Behavioral Therapy; Ethanol

STUDY DESIGN:
Intervention Model Description: In addition to Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT-AUD), participants will be randomized to receive sleep education or to participate in 5 individual sessions of Cognitive Behavioral Therapy for Insomnia (CBT-I).
Who Masked: Participant, Outcomes Assessor
Masking Description: The project manager will inform study therapists of participant assignment to conditions. PI Miller and study therapists will be blinded to assessment outcomes, and the assessment RA will be blinded to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I + AUD-TAU (Experimental): Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week for five (5) weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Alcohol Use Disorder Treatment as Usual
- Sleep Hygiene + AUD-TAU (Active Comparator): Sleep hygiene education delivered once to all participants
  Interventions: Behavioral: Sleep Hygiene; Behavioral: Alcohol Use Disorder Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Study therapists will follow the 2014 CBT-I in Veterans manual developed by leading researchers in the behavioral sleep medicine field. Intervention components include (1) sleep hygiene: limiting naps; avoiding caffeine, tobacco, alcohol, and rich/heavy foods before bedtime; exercising; establishing a bedtime routine; and creating a comfortable sleep environment; (2) sleep restriction: limiting time in bed in order to improve sleep efficiency, or the percentage of time in bed that is actually spent sleeping; time in bed will be titrated each week based on sleep efficiency; (3) stimulus control: strengthening association between bedroom and sleep to decrease conditioned arousal; (4) relaxation: diaphragmatic breathing, progressive muscle relaxation, and visual imagery to reduce arousal; and (5) cognitive therapy: identifying and challenging thoughts that interfere with sleep.
  Arms: CBT-I + AUD-TAU
Behavioral: Sleep Hygiene — Study therapists will review a one-page handout on sleep hygiene with all participants. This is the only intervention that participants assigned to the sleep hygiene condition will receive. This is consistent with what may be expected as standard care in a doctor's visit with a primary care physician.
  Arms: Sleep Hygiene + AUD-TAU
Behavioral: Alcohol Use Disorder Treatment as Usual — CBT-based groups for Alcohol Use Disorder will focus on the acquisition of skills needed to cope effectively with urges and cravings to drink and manage high-risk situations.
  Other Names: AUD-TAU

SUMMARY:
Project SAVE aims to examine the feasibility, acceptability, and initial efficacy of a CBT-I supplement to alcohol treatment of Veterans.

DETAILED DESCRIPTION:
Alcohol use disorders (AUDs) are prevalent among Veterans and result in significant physical and psychological burden. Among those who receive treatment for AUDs, 1 in 3 relapses to problematic drinking within one year of treatment. Thus, additional strategies are needed to enhance alcohol treatment outcomes. One promising approach involves providing concurrent treatment for a common complaint - difficulty falling or staying asleep. Up to 74% of Veterans seeking treatment for AUD report co-occurring symptoms of insomnia. Given the negative impact of insomnia on attention and emotion regulation, insomnia symptoms may decrease patients' abilities to attend to alcohol treatment and manage negative emotions that lead to craving and relapse. Moreover, approximately 50% of individuals with AUDs report using alcohol to help them sleep, making relapse more likely for those with no other tools or skills to help them sleep. Indeed, sleep disturbance has been identified as a risk factor for relapse among individuals in alcohol treatment. Thus, effective treatment of sleep problems may enhance alcohol treatment. Cognitive Behavioral Therapy for Insomnia (CBT-I) has been effective in reducing insomnia severity in individuals with AUDs; however, no investigations have examined the efficacy of CBT-I delivered concurrently with AUD treatment to determine its impact on treatment outcomes. This R21 aims to examine the feasibility, acceptability, and initial efficacy of a CBT-I supplement to ongoing alcohol treatment. A randomized pilot trial with 80 Veterans who meet diagnostic criteria for AUD and Insomnia Disorder will be conducted. Participants will be randomly assigned to receive Cognitive Behavioral Therapy for Insomnia (CBT-I) or minimal treatment (educational handout only; EDU) in addition to alcohol treatment as usual. Outcomes will be assessed at the end of the active intervention period (6 weeks) and 6 weeks post-intervention. Preliminary process outcomes include recruitment/retention rates and treatment satisfaction (feasibility and acceptability, respectively). Primary outcomes are insomnia severity, percentage of heavy drinking days, and alcohol-related problems; and we plan to examine post-treatment changes in insomnia severity as a mediator of treatment effects on alcohol use outcomes. We will also assess treatment effects on a variety of secondary clinical and mechanistic outcomes (e.g., PTSD symptoms, attention, working memory, treatment-related learning). Multiple imputation will be used for missing data, and analyses will be intent-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Participation in alcohol treatment at the Truman VA (Columbia, MO)
* DSM-5 criteria for moderate to severe Alcohol Use Disorder
* Substance use in the past 2 months
* DSM-5 episodic criterion (duration at least 1 month) for Insomnia Disorder

Exclusion Criteria:

* unable to provide informed consent
* cognitive impairment
* continuous sobriety for 2+ months at baseline
* manic episode or seizure in the past year (contraindications for CBT-I)
* severe psychiatric disorder that requires immediate clinical attention
* initiation of a sleep medication in the past six (6) weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Miller, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the research team to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared after data collection is complete and results have been published (anticipated July 2022).
Access Criteria: De-identified data will be made available to other qualified investigators who aim to verify data, conduct meta-analyses, or collaborate with the research team on analyses that are not already planned.

REFERENCES:
- [Derived] Miller MB, Carpenter RW, Freeman LK, Dunsiger S, McGeary JE, Borsari B, McCrae CS, Arnedt JT, Korte P, Merrill JE, Carey KB, Metrik J. Effect of Cognitive Behavioral Therapy for Insomnia on Alcohol Treatment Outcomes Among US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Sep 1;80(9):905-913. doi: 10.1001/jamapsychiatry.2023.1971. PMID 37342036
- [Derived] Miller MB, Metrik J, McGeary JE, Borsari B, McCrae CS, Maddoux J, Arnedt JT, Merrill JE, Carey KB. Protocol for the Project SAVE randomised controlled trial examining CBT for insomnia among veterans in treatment for alcohol use disorder. BMJ Open. 2021 Jun 8;11(6):e045667. doi: 10.1136/bmjopen-2020-045667. PMID 34103317

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Started | 32 | 35
Completed | 28 | 35
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.9) | 46.9 (11.9) | 46.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 29 | 32 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Multiracial or multiethnic | 4 | 0 | 4
  Race/ethnicity: White only | 26 | 30 | 56
  Race/ethnicity: Black or African American | 1 | 5 | 6
  Race/ethnicity: Hispanic or Latinx | 1 | 0 | 1
Highest level of education [Count of Participants; unit: Participants]
  Some high school | 1 | 0 | 1
  High school graduate or GED | 6 | 7 | 13
  Some college | 16 | 18 | 34
  College graduate | 9 | 10 | 19
Housing [Count of Participants; unit: Participants]
  My own house/apt | 20 | 16 | 36
  Someone else's house/apt | 7 | 5 | 12
  Transitional/institutional housing | 5 | 11 | 16
  On the street | 0 | 3 | 3
Marital status [Count of Participants; unit: Participants]
  Never married | 6 | 4 | 10
  Married or living with partner | 11 | 8 | 19
  Divorced, separated, widowed | 15 | 23 | 38
Branch [Count of Participants; unit: Participants]
  Air Force | 4 | 3 | 7
  Army | 22 | 21 | 43
  Marines | 2 | 5 | 7
  Navy | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity
Description: Assessed using the Insomnia Severity Index (ISI); ISI will be used as a 7-item measure of insomnia severity in the past two weeks. Items assess difficulty falling or staying asleep, satisfaction with current sleep pattern, interference with daily functioning, the extent to which others notice their sleep problems, and worry/distress related to sleep problems. Response options for each item range from 0 (not at all worried) to 4 (very much worried). Individual item scores are summed to a total score - the highest possible score being 28. Higher scores indicate more severe insomnia. Participants scoring 10 or higher will be classified as screening positive for insomnia.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 17.97 (4.66) | 19.26 (4.01)
  6 weeks | 5.69 (4.70) | 10.96 (6.43)
  12 weeks | 8.07 (7.13) | 12.42 (6.34)

2. Primary Outcome: Percent of Heavy-drinking Days
Description: Assessed using the Timeline Followback (TLFB) for alcohol; TLFB allows participants to trace their alcohol use back 30 days.
Time Frame: Baseline to post-treatment (week 6) to follow-up (week 12)
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
percentage of heavy drinking days
  Baseline | 16.97 (9.58) | 17.14 (11.74)
  6 weeks | 2.07 (5.26) | 1.34 (4.49)
  12 weeks | 5.92 (11.45) | 6.57 (13.56)

3. Primary Outcome: Alcohol Problems
Description: Assessed using the Short Inventory of Problems (SIP). SIP measures adverse consequences of substance use. Scores range 0 to 45, where higher scores indicate more frequent problems.
Time Frame: Baseline to post-treatment (week 6) to follow-up (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 25.44 (10.11) | 22.00 (12.17)
  6 weeks | 4.42 (6.19) | 5.12 (9.10)
  12 weeks | 4.38 (7.65) | 7.00 (9.03)

4. Secondary Outcome: Sleep Efficiency
Description: Assessed using daily sleep diaries. Sleep Diaries are quotidian questionnaires that measure self-reported sleep quality, sleep & wake time, and daily habits concerning substance use. Scores range 0 to 100, where higher scores indicate better (more favorable) sleep efficiency. Treatment goal is 85%.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
percentage
  Baseline | 68.47 (11.91) | 71.44 (13.32)
  6 weeks | 87.30 (7.50) | 82.41 (11.51)
  12 weeks | 90.62 (5.26) | 75.31 (14.11)

5. Secondary Outcome: Post-Traumatic Stress Disorder Symptoms
Description: Assessed using the Post-Traumatic Stress Disorder Checklist from the Diagnostic and Statistical Manual-5 (PCL-5); PCL-5 is a 20-item measure of Post-Traumatic Stress Disorder (PTSD). On a scale of not at all (0) to extremely (4), participants indicate how frequently in the past month they were bothered by stressful experiences such as disturbing dreams, hyper-alertness, strong negative beliefs, and irritability. PCL-5 is scored by summing the responses. Possible scores range from 0-80, where higher scores indicate higher PTSD severity.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CBT-I: 5-session cognitive behavioral therapy for insomnia
- Sleep Hygiene: single session of sleep hygiene recommendations
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 34.3 (22.3) | 32.0 (21.6)
  6 weeks | 20.1 (21.1) | 25.2 (22.1)
  12 weeks | 21.0 (22.1) | 28.2 (24.8)

6. Secondary Outcome: Symptoms of Depression
Description: Assessed using the Patient Health Questionnaire-9 (PHQ-9); PHQ-9 will be used as a 9-item measure of depressed mood and functioning that has demonstrated good sensitivity and specificity across adult samples. Participants will indicate how many days in the past two weeks (not at all, several days, more than half the days, or every day or nearly every day) they have experienced each problem. Scores range from 0 to 27, where higher scores indicate more severe symptoms of depression.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Population: Some participants lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 10.9 (5.6) | 12.3 (5.6)
  6 weeks: number analyzed (Participants) | 26 | 26
  6 weeks | 4.7 (4.7) | 7.4 (6.3)
  12 weeks: number analyzed (Participants) | 27 | 24
  12 weeks | 7.3 (6.0) | 8.9 (7.5)

7. Secondary Outcome: Symptoms of Anxiety
Description: Assessed using the Generalized Anxiety Disorder-7 (GAD-7); GAD-7 is a 7-item measure of anxiety with strong criterion and predictive validity. On a scale from not at all (0) to nearly every day (3), participants indicate how often in the past two weeks they have experienced problems such as having trouble relaxing and being so restless that it is hard to sit still. Possible total scores range from 0-21. Scores will be summed and classified as minimal anxiety (<3), moderate anxiety (4-7), high anxiety (12-15), or severe anxiety (16-21).
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Population: Some participants lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 9.8 (10.8) | 10.8 (5.8)
  6 weeks: number analyzed (Participants) | 26 | 26
  6 weeks | 4.9 (4.3) | 7.0 (5.7)
  12 weeks: number analyzed (Participants) | 27 | 24
  12 weeks | 7.2 (6.6) | 8.7 (5.6)

8. Secondary Outcome: Treatment-Related Learning
Description: Assessed using the Project SAVE alcohol quiz
Time Frame: Change from baseline to post-treatment (week 6)
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Days Where Alcohol Was Used to Help With Sleep
Description: Assessed using the daily sleep diary; Did you use alcohol specifically to help with sleep?
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
percentage of days
  Baseline | 3.68 (16.86) | 2.94 (14.83)
  6 weeks | 4.08 (15.48) | 4.76 (21.82)
  12 weeks | 8.09 (18.55) | 3.16 (8.44)

10. Secondary Outcome: Alcohol Craving
Description: Assessed using the Penn Alcohol Craving Scale (PACS); The Penn Alcohol Craving Scale is a 5-item measure of alcohol craving in the past week. Participants rate the intensity, frequency, and duration of cravings, as well as their ability to resist acting on those cravings and their overall "average alcohol craving" for the past week. This measure has demonstrated good internal consistency and construct validity. Scores range 0 to 30, where higher scores indicate stronger craving.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 11.44 (8.85) | 10.76 (7.59)
  6 weeks | 7.88 (6.73) | 7.15 (6.25)
  12 weeks | 9.31 (7.25) | 9.21 (6.86)

11. Secondary Outcome: Negative Affect
Description: Assessed using the Positive and Negative Affect Schedule (PANAS); Negative affect subscale scores range from 10-50, with higher scores indicating more extreme negative affect (measured "right now").
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Population: Some participants lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 35 | 32
score on a scale
  Baseline | 20.0 (8.7) | 20.3 (9.0)
  6 weeks: number analyzed (Participants) | 26 | 26
  6 weeks | 15.2 (4.5) | 16.5 (7.5)
  12 weeks: number analyzed (Participants) | 27 | 24
  12 weeks | 18.2 (7.8) | 20.0 (10.6)

12. Secondary Outcome: Emotion Regulation
Description: Assessed using the Brief Difficulties in Emotion Regulation Scale (DERS-16). The 16-item Difficulties in Emotion Regulation Scale has demonstrated good convergent and discriminant validity in clinical and community samples (Bjureberg et al., 2015). Scores range from 16 to 80, with higher scores indicating more difficulties with emotion regulation.
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Population: Some participants lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 32 | 35
score on a scale
  Baseline | 20.0 (8.7) | 20.3 (9.0)
  6 weeks: number analyzed (Participants) | 26 | 26
  6 weeks | 15.2 (4.5) | 18.2 (7.8)
  12 weeks: number analyzed (Participants) | 27 | 24
  12 weeks | 18.2 (7.8) | 20.0 (10.6)

13. Secondary Outcome: Delay Discounting
Description: Assessed using the Monetary Choice Questionnaire (MCQ); The MCQ (Kirby, Petry, & Bickel, 1999) will be used as a self-report measure of delay discounting. In 27 trials, participants will be asked to choose between a smaller, immediate reward or a larger, delayed reward. For example, "Would you prefer $54 today or $55 in 117 days?" Data will be used to calculate participants' discounting-rate parameter (k).
Time Frame: Baseline to post-treatment (week 6) to follow up (week 12)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CBT-I + AUD-TAU | Sleep Hygiene + AUD-TAU
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03806491/Prot_SAP_000.pdf